CLINICAL TRIAL: NCT02752581
Title: Efficacy of Peroperative Suction Drain Usage in Arthroscopic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mert Özcan (Other)
Responsible Party: Sponsor-Investigator, Mert Özcan, Assoc. Prof., Trakya University
Organization: Trakya University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TÜTFEK 2008/201
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Chondropathy; Knee Effusion; Knee Hemarthrosis
Keywords: suction drain; knee arthroscopy; knee pain
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drain Group (Other): Suction drain was applied to these patients after arthroscopic knee surgery.
  Interventions: Device: Suction drain
- Control Group (Other): No suction drain was applied to this group, therefore used as a control group.
  Interventions: Device: No suction drain

INTERVENTIONS:
Device: Suction drain — A suction drain is used to remove excess fluid from tissues after surgery.
  Other Names: Hemovac drain
  Arms: Drain Group
Device: No suction drain — A suction drain is used to remove excess fluid from tissues after surgery.
  Arms: Control Group

SUMMARY:
The study was designed to investigate efficacy of suction drains in arthroscopic knee surgery, rather than anterior cruciate ligament (ACL) reconstruction. two groups were randomised, and suction drain was applied to one group, and the other group as the control group without a suction drain.

DETAILED DESCRIPTION:
The groups were compared in terms of patellar shock, knee effusion, knee scoring systems, range of motion, loss of labour, hospitalization time. Also different arthroscopic procedures such as meniscectomy, meniscus repair, synovectomy and microfracture were evaluated in terms of need for a suction drain. The controls was at 1st and 15th day, 6th week and 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee derangement and accepted to enroll to the study

Exclusion Criteria:

* intraarticular fracture, ACL surgery, arthrotomy, bleeding disorder,

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Activity Pain | 3 months
  Severity of pain was evaluated with Visual Analogue Scale (VAS). VAS is a horizontal line divided into ten equal intervals in which zero represents no pain and 10 represents the worst pain ever felt.
Rest Pain | 3 months
  Severity of pain was evaluated with Visual Analogue Scale (VAS). VAS is a horizontal line divided into ten equal intervals in which zero represents no pain and 10 represents the worst pain ever felt.
Range of Motion | 3 months
  Range of motion is measures in terms of angular degrees.

SECONDARY OUTCOMES:
Lysholm | 3 months
  Lysholm is a scoring system from zero to one hundred. It measures subjective complaints of the patients.
International Knee Documentation Committee Score | 3 months
  is a scoring system from zero to one hundred. It measures subjective complaints of the patients.
hospitalization time | 1 month
  It is measured in days. It shows the period of hospitalization time, from surgery to discharge.
loss of labour time | 1 month
  It is measured in days. It shows the time from discharge to beginning of work.

OTHER OUTCOMES:
Amount of drainage | 1 day
  The amount of fluid in suction drain. It is measured with cubic centimetre (cc).
patellar shock | 1.5 months
  Patellar shock was graded in four scales: Grade 1, some notable fluid, Grade 2, minimally elevated patella, Grade 3, patellar ballottement, and Grade 4, tense knee capsule, unable to compress patella.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Browett JP, Gibbs AN, Copeland SA, Deliss LJ. The use of suction drainage in the operation of meniscectomy. J Bone Joint Surg Br. 1978 Nov;60-B(4):516-9. doi: 10.1302/0301-620X.60B4.711799.
- [Background] Alkan K, Unay K, Berkem L, Guven M, Poyanli O. Suction drainage influence on knee effusion following partial meniscectomy with partial fat pad or synovium resection. Acta Orthop Traumatol Turc. 2011;45(4):221-4. doi: 10.3944/AOTT.2011.2545. PMID 21908960
- [Background] Tatari H, Dervisbey M, Muratli K, Ergor A. Report of experience in 190 patients with the use of closed suction drainage in arthroscopic knee procedures. Knee Surg Sports Traumatol Arthrosc. 2005 Sep;13(6):458-62. doi: 10.1007/s00167-004-0537-1. Epub 2004 Nov 13. PMID 16170580